CLINICAL TRIAL: NCT05130398
Title: A Phase 1/2, Randomized, Controlled Open-label Trial to Evaluate the Safety and Immunogenicity of the rVSVΔG-ZEBOV-GP Ebola Virus Vaccine Candidate in Healthy Children Aged 1 to 12 Years and in Their Relatives Living in Lambaréné, Gabon
Brief Title: Safety and Immunogenicity of the rVSVΔG-ZEBOV-GP Ebola Virus Vaccine Candidate in Children Living in Lambaréné, Gabon
Acronym: EBOLAPED
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre de Recherche Médicale de Lambaréné (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Selidji Todagbe Todagbe Agnandji, Director, Centre de Recherche Médicale de Lambaréné
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LA rVSVΔG-ZEBOV-GP -02-PED
Record Dates: First submitted 2021-08-25; First posted 2021-11-23 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Ebola Virus Disease
Keywords: Sub-Saharan Africa Africa ,; Children; rVSV-ZEBOV-GP vaccine; Shedding; Safety; Tolerability
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — Dietary Fiber; Lunch; Chickenpox Vaccine

STUDY DESIGN:
Intervention Model Description: A Phase 1/2, randomized, controlled, open label clinical trial.
Masking Description: The vaccine doses of ≥7.8 x 107 pfu will be evaluated and compared to vaccination with varicella vaccine as a control. In addition, the closest contact persons of the vaccinees will be monitored for possible transmission of the viral vaccine vector.
  The study will enroll children of two age groups living in Lambaréné, Gabon. Children will be followed-up for 12 months post vaccination.
  The 1-2 closest contact persons of each participant will be involved in the monitoring of rVSV transmission.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- the rVSVΔG-ZEBOV-GP vaccine (Experimental): Participants of the experimental arm will receive a single intramuscular dose of ≥7.8 x 107 pfu of the rVSVΔG-ZEBOV-GP vaccine. In total, 80 participants will receive the experimental vaccine: 40 participants aged 6-12 years and 40 aged 1-5 years.
  Interventions: Biological: rVSVΔG-ZEBOV-GP, V920
- The Chikenpox or Varicella (Varilix) vaccine (Active Comparator): The control arm consists of the chickenpox vaccine. Forty children will receive a single subcutaneous dose of Varilix, the active comparator vaccine, 20 aged 6-12 years and 20 aged 1-5 years
  Interventions: Biological: Chikenpox or Varicella vaccine (VARILRIX)
- Fibre and equilibrate diet (Experimental): Participants were assigned to receive two meals daily ( breakfast and lunch) for 21 days. About 30 children are randomly assigned to fibre and equilibrate diet.
  Interventions: Dietary Supplement: Fibre and equilibrate breakfast and lunch
- Active detection and treatment of pathogens according to standard of care (Experimental): The following pathogens: P. falciparum, Ascaris lumbricoides, Trichuris trichiura, Necator americanus, intestinal protozoa, BG+, BG- colonies and pathogens, SARS-CoV2 are actively detected and treated according to the standard of care every month. About 30 children are randomly assigned to this arm.
  Interventions: Diagnostic Test: Active detection and treatment of pathogens
- Diet plus Active detection and treatment of pathogens according to standard of care (Experimental): Participants were assigned to receive two meals daily ( breakfast and lunch) for 21 days and concomitantly assigned to active detection of P. falciparum, Ascaris lumbricoides, Trichuris trichiura, Necator americanus, intestinal protozoa, BG+, BG- colonies and pathogens, SARS-CoV2 every month. About 30 children are assigned to receive combined interventions
  Interventions: Combination Product: Fibre and equilibrate breakfast and lunch plus Active detection and treatment of pathogens
- No diet and no pathogen detection (Placebo Comparator): About 30 children received no diet and no active detection of pathogens
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: rVSVΔG-ZEBOV-GP, V920 — The experimental vaccine is the rVSVΔG-ZEBOV-GP, an Ebola vaccine.
  Arms: the rVSVΔG-ZEBOV-GP vaccine
Dietary Supplement: Fibre and equilibrate breakfast and lunch — Participants receive fibres and caloric equilibrate diet during breakfast and lunch every day for 21 consecutive days.
  Arms: Fibre and equilibrate diet
Diagnostic Test: Active detection and treatment of pathogens — Monthly diagnostic and treatment of childhood infections Active detection and treatment of pathogens.
  Arms: Active detection and treatment of pathogens according to standard of care
Combination Product: Fibre and equilibrate breakfast and lunch plus Active detection and treatment of pathogens — Participants receive fibres and caloric equilibrate diet during breakfast and lunch every day for 21 consecutive days and diagnostic and treatment of childhood infections Active detection and treatment of pathogens every month for 12 months
  Arms: Diet plus Active detection and treatment of pathogens according to standard of care
Biological: Chikenpox or Varicella vaccine (VARILRIX) — The active comparator vaccine, a Varicella vaccine (VARILRIX®)
  Arms: The Chikenpox or Varicella (Varilix) vaccine
Other: Placebo — About 30 children do not receive diet, nor active pathogen detection
  Arms: No diet and no pathogen detection

SUMMARY:
LA rVSVΔG-ZEBOV-GP -02-PED is a Phase 1/2, randomized, controlled open label trial. The LA rVSVΔG-ZEBOV-GP -02-PED trial aims primarily to assess the clinical significance of shedding of the rVSV RNA following vaccination with the rVSVΔG-ZEBOV-GP vaccine in children. The vaccine doses of ≥7.8 x 107 pfu will be evaluated and compared to vaccination with varicella vaccine as a control. In addition, the closest contact persons of the vaccinees will be monitored for possible transmission of the viral vaccine vector.

The study will enroll children of two age groups living in Lambaréné, Gabon. Children will be followed-up for 12 months post vaccination.

The 1-2 closest contact persons of each participant will be involved in the monitoring of rVSV transmission. They will be followed until day 56 post- vaccination of their children/ sibling.

DETAILED DESCRIPTION:
LA-rVSVΔG-ZEBOV-GP -02-PED is a Phase 1/2, randomized, controlled, open label, trial and is designed to generate further safety, tolerability and immunogenicity data of the 7.8 x 107 PFU rVSVΔG-ZEBOV-GP vaccine in children aged 1 -12 years living in a sub-Saharan Africa. The study will enroll participants into two age groups. A total of 120 children will be enrolled and followed-up for 12 months post injection. In addition, a maximum of 240 relatives of the study participants will be enrolled to assess the transmission of the rVSVΔG-ZEBOV-GP vaccine.

Group 1: 60 participants aged 6-12 years will be randomized in group 1. 40 participants will receive a single intramuscular dose of 7.8 x 107 pfu rVSVΔG-ZEBOV-GP vaccine. 20 participants will receive a single subcutaneous dose of varicella vaccine The participants will be allocated to each treatment at a ratio of 2:1 respectively Group 2: 60 participants aged 1 -5 years will be randomized into group 2. 40 will receive a single intramuscular dose of 7.8 x 107 pfu of rVSV-ZEBOV vaccine. 20 participants will receive a single subcutaneous dose of varicella vaccine The participants will be allocated to each treatment at a ratio of 2:1 respectively

Vaccinations will start in group 2 after the first 10 participants of group 1 have completed the day 28 post vaccination visit and the SMC has done a review of safety data until that point.

For each vaccinee there will be a 365 -day period of follow-up after vaccination. The contact persons of the vaccinees will be followed-up until day 56 after the vaccination of their relative.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 1 to 12 years (inclusive) at the time of inclusion.
* Willingness of parent or legal guardian to provide written informed consent prior to screening procedures.
* Willingness of the relatives of the participant to provide written informed consent if they are ≥ 18 years (or an assent when they are 13 to 17 years old).
* Available, able, and willing to participate in all study visits and procedures

Exclusion Criteria:

* History of severe local or systemic reactions to any vaccination or a history of severe allergic reactions, or known allergy to the components of the vaccines.
* Ongoing participation in another clinical trial
* Participation in previous Ebola vaccine trials
* Receipt of a licensed vaccine within 14 days of planned study immunization (30 days for live vaccines)
* Presence of any febrile illness (fever >38°C) or any moderate to severe illness within one week prior to vaccination;
* Administration of immunoglobulins and/or any blood products within the 120 days preceding study entry or planned administration during the study period
* Any other significant finding that in the opinion of the investigator would increase the risk of the individual having an adverse outcome from participating in this study.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Concentration of viral vector in blood, saliva and urine in vaccinees | at days 0, 1, 2/3, 7, 14 and 28
  Concentration of rVSVΔG-ZEBOV-GP in blood, urine, or saliva as detected by RT-PCR and expressed as copy number in vaccinees
Prevalence and relative risk of sollicited adverse events in vaccinees | until day 14 post vaccination
  Proportion (percent) of participants experiencing sollicited adverse events in vaccinees groups
Prevalence and relative risk of unsolicited adverse events and serious adverse events in vaccinees | until day 28 after vaccination
  Proportion (percent ) of participant experiencing unsollicited adverse event (AEs) and serious adverse events (SAEs) and relative risk of AEs and SAEs in participant by vaccine groups

SECONDARY OUTCOMES:
Prevalence and relative risk of serious adverse events | until day 365
  Proportion (percent) of participants experiencing SAEs and relative risk of SAEs in until study last visit (at 365 days)
Transmission intensity of the viral vector in blood, saliva and urine among the the relatives of the vaccinees | days 0, 1, 3, 14, 28, 56
  Concentration of rVSVΔG-ZEBOV-GP in blood, urine, or saliva as detected by RT-PCR and expressed as copy number in the close relatives of the vaccinees
Titres of ZEBOV-GP-specific binding antibody | days 0, 1, 3, 14, 21, 28, 56, 84, 180, 365
  Titres of ZEBOV-GP-specific binding antibody by ELISA expressed in geometric mean titres (GMTs)
Affinity/Avidity of antibody induced by vaccination | days 28 and 180
  Affinity/avidity of GP-specific serum antibodies as assessed by Surface Plasmon Resonance platform at D28 and D180 expressed as percent of affinity maturation
Concentration of IL-1RN (IL-1Ra), IL-6, TNF-α, IL-10, MCP-1/CCL2, and MIP-1β/CCL4 | days 0, 1 and 2 or 3
  Cytokines (IL-1RN (IL-1Ra), IL-6, TNF-α, IL-10), chemokines and soluble adhesion molecules (MCP-1/CCL2, and MIP-1β/CCL4) plasma expressed in microgram per milliliter .
Prevalence of miRNAs | at days 0, 1, 2/3, 7
  Proportion (percent) of circulating miRNAs using the Human miRNome PCR array v.21 in serum samples
Concentration of Lipids, glutamine, Alanine, Aspargine | at day 0, day 1, day 2/3 and day 7
  Proportion (percent ) and concentration ( microgram/ mililiter) of Lipids, glutamine, Alanine, Aspargine in plasma samples
Concentrations Nitric oxides species | days 0, 1, 2/3, 7, 28, 56, 90, 180, 365
  Profiling nitric oxides species according to vaccines, diet and pathogens
Concentration of metabolites of gut bacteria | days 0, 7, 28, 56, 90
  Measurement of gut metabolites
Titres of antibody induced by diphtheria, tetanus, Bordetella, poliomyelitis, hepatitis B, measles, yellow fever ( EPI vaccines) | days 0, 7, 14, 28, 90, 180, 365
  Concentration of antibody of EPI vaccines
Concentration of bystander cytokines | days 0, 1, 2/3, 7, 28, 90
  Concentration of cytokines that may induce heterologous vaccine induced immune responses

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherches Médicales de Lambaréné, Lambaréné, Moyen-Ogooué Province, Gabon

IPD SHARING:
Plan to Share IPD: Yes
The Principal investigator or his designee will be the data manager with responsibility for delegating the receiving, entering, cleaning, querying, analysing and storing all data that accrues from the study. All data will be entered in paper case record forms and transcribed by double entry into an electronic database. This includes safety data, laboratory data (both clinical and immunological) and outcome data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From preliminary intererim analysis until the final report fo the study.The site owns the data and it is agreed that publication will occur in a timely manner.
Access Criteria: All files and source documents will be kept confidentially in locked safety cabinets. The Principal investigator, co-investigators and clinical research nurses will have access to records. The investigators will permit authorized representatives of the sponsor, regulatory agencies and the monitors to examine (and when required by applicable law, to copy) clinical records for the purposes of quality assurance reviews, audits and evaluation of the study safety and progress.